CLINICAL TRIAL: NCT06626386
Title: Determination of Prostate-specific Antigen in Capillary Blood (PSA-Cap)
Acronym: PSA-Cap
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Rouvier Al-Monajjed, Oberarzt, Heinrich-Heine University, Duesseldorf
Other Study IDs: 006
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate specific Antigen
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PSA testing — PSA Testing in venipunctate and capillary blood

SUMMARY:
The aim of the PSA-Cap study is to test the comparability of measurements of total PSA in serum from venipuncture and in serum from capillary blood using anonymized diagnostic blood samples from patients. Furthermore, a stability test of the samples is carried out after storage at room temperature for 24, 72/96 and 168 hours. Particular attention is paid to the comparability of the measurement results and the influence of the transportation time.

DETAILED DESCRIPTION:
Interventions that are conducted with the PSA-Cap trial are the collection of capillary blood (6 droplets) from the fingertip during regular PSA testing in venous blood. PSA is measured in the serum fraction of both samples (capillary and venous) using the established routine procedure, either immediately or after simulation of common transport conditions (intermediate storage for 24; 72/96 h and 168 h at 22 °C). Control measurements include parameters of cell lysis (LDH, HIL check) and general protein stability (albumin). The patient samples used are anonymized at the source by means of a consecutive series of numbers. The anonymized result groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Men aged from 45 to 70 years
* Informed consent for PSA measurement for prostate cancer screening

Exclusion Criteria:

* Patients unable to give consent

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients between the ages of 40 and 70 who receive a PSA test as part of their routine examination
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of PSA measurement in capillary blood vs. venous blood | After 0 h, 1 d, 3/4 d and 7 d

SECONDARY OUTCOMES:
PSA stability in serum fraction of both samples (capillary and venous) | After 0 h, 1 d, 3/4 d and 7 d

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Urologie, Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No